CLINICAL TRIAL: NCT01802359
Title: Post-Marketing Surveillance of Bravonto in Korea
Brief Title: A Study to Evaluate the Safety and Effectiveness of Mirodenafil in Korean Patients With Erectile Dysfunction
Status: Terminated | Type: Observational
Why Stopped: This prodect will be transferred to another company.
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100836; MIRODENEDY4002 (Other: Janssen Korea, Ltd., Korea); MIR-KOR-PMS (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2013-02-28; First posted 2013-03-01 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Mirodenafil; Bravonto
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mirodenafil
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Korean male participants receiving mirodenafil as per the prescribing information will be observed.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of mirodenafil in participants with erectile dysfunction.

DETAILED DESCRIPTION:
This is a non randomized (the study medication is not assigned by chance), open-label (all participants and study staff know the identity of the treatment), multi-center, prospective (looking forward using observations collected following participant enrollment), and non-comparative study in which participants with erectile dysfunction will be observed to evaluate the safety and effectiveness of mirodenafil for 12 weeks. Safety evaluations will include assessment of adverse events, and record of concomitant medications. The study will be conducted in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with erectile dysfunction
* Participants prescribed mirodenafil on demand

Exclusion Criteria:

- Participants who have administered mirodenafil for other than an approved indication

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with erectile dysfunction and prescribed mirodenafil on demand.
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2011-11-07 (Actual); Primary Completion 2012-05-31 (Actual); Study Completion 2012-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 4 weeks

SECONDARY OUTCOMES:
International Index of Erectile Function | Baseline (Week 0), Week 4, Week 8, and Week 12
  The International Index of Erectile Function is used for the assessment of erectile dysfunction, with scores ranging from 0 to 30. Evaluation of points are as follows: 1-10 = severe erectile dysfunction, 11-16 = moderate dysfunction, 17-21 = mild to moderate dysfunction, 22-25 = mild dysfunction, 26-30 = no dysfunction. Lower scores indicate worsening.
Sexual Encounter Profile | Baseline (Week 0), Week 4, Week 8, and Week 12
  The Sexual Encounter Profile is assessed after each sexual attempt consisting of a series of yes/no questions regarding specific aspects of each encounter. Question 1 asks, "Were you able to insert your penis into your partner's vagina?" and question 2 asks, "Did your erection last long enough for you to complete intercourse with ejaculation?".
Global assessment Questionnaire | Baseline (Week 0), Week 4, Week 8, and Week 12
  The Global Assessment Questionnaire is a self-administered questionnaire (Yes/No) that allows men to rate improvement in erectile function. Question 1 asks "Has the treatment you have been taking over the past 4 weeks improved your erections?" and if the answer is yes, question 2 then asks "Has the treatment improved your ability to engage in sexual activity"
Number of participants with adverse events | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea